CLINICAL TRIAL: NCT06734845
Title: Energy Status and Protein Intake As Prognostic Indicators of Rehabilitative Outcomes
Acronym: ESPI-PRO
Status: Completed | Type: Observational
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Nancy Rodriguez, Professor Emerita, University of Connecticut
Other Study IDs: HHC-2022-0261
Record Dates: First submitted 2024-03-18; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Orthopedic; Osteo Arthritis Knee; Hip Osteoarthritis; Protein-Energy Malnutrition; Energy Malnutrition Protein
Keywords: Joint replacement; Rehabilitation; Protein; Energy Balance; Knee arthroplasty; Hip arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Protein-Energy Malnutrition; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Total Knee Arthroplasty: Patients undergoing first total knee replacement
  Interventions: Procedure: Total Knee Arthroplasty
- Total Hip Arthroplasty: Patients undergoing first total hip replacement
  Interventions: Procedure: Total Joint Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total Joint (Knee or Hip) Arthroplasty
  Other Names: Total Hip Arthroplasty
  Groups: Total Knee Arthroplasty
Procedure: Total Joint Arthroplasty — Participants will be patients undergoing first total knee or total hip replacement
  Groups: Total Hip Arthroplasty

SUMMARY:
The proposed project is novel in its goal to establish a foundation for evidence-based rehabilitative nutrition guidelines to enhance perioperative patient care and improve post-operative rehabilitative outcomes specific to muscle health (muscle mass, strength, and function) and quality of life in elective orthopedic surgery patients undergoing total joint replacement procedures.

Study Aims. Specific aims and their respective approach for the proposed investigation were:

Aim 1: Characterize energy status and protein intake in total hip arthroplasty and total knee arthroplasty patients prior to surgery.

Approach. Following approval of investigation by the Hartford Hospital Institution Review Board, data collection involved the inclusion of a research information sheet and a 3-day food record with instructions for the respective patient to complete prior to surgery.

Aim 2: Evaluate association between energy status, positive or negative energy balance on standard outcome measures assessed throughout physical rehabilitation to determine whether energy status and protein intake at admission predicts objective and subjective rehabilitative outcome measures. Dietary assessments (3-day food record, protein screener) occurred at time points corresponding to physical rehabilitative assessments per approach for Aim 1.

Approach. Total Hip Replacement assessments will occur between Day 1 following surgery and Week 2 and 6 months post surgery . Outcome measures included Pain Visual Analog Scale, Hip Disability Osteoarthritis Outcome Score, Timed Up and Go Test, 30 second Sit to Stand Test, Passive Hip Range of Motion and Active Hip Range of Motion.

Total knee assessments were taken post surgery on between Day 1 and Week 2 and at 4 to 6 Weeks, and 7 to 12 Weeks following surgery. These included Pain Visual Analog Scale, Knee Injury and Osteoarthritis Outcome Score, Timed Up and Go test, 30-second Sit to Stand Test, Passive and Active Knee Range of Motion, and Knee Strength.

Aim 3: Validate a protein screener developed by our research team and designed to characterize protein intake and protein source was administered pre- and post-operatively.

For the latter, time points were established according to respective treatment guidelines for Total Hip and Total Knee replacement patients, respectively.

DETAILED DESCRIPTION:
Clinical Significance: The clinical relevance of the proposed project is the eventual development of evidence-based rehabilitative nutrition practice guidelines for orthopedic patients. The scientific literature specific to the role of perioperative nutrition on rehabilitative outcomes in patients undergoing elective total joint procedures, total hip arthroplasty and total knee arthroplasty in particular, is limited.

Background and Study Rationale. Orthopedic procedures are commonly undergone to treat injuries and chronic conditions affecting the hip and knee. Primary arthroplasties represented 86% of the 1.9 million hip and knee arthroplasties performed in the United States from 2012-2019. Total hip and total knee replacement procedures are typical in older men and women and persistent muscle loss is a shared clinical presentation for young as well as older individuals undergoing elective orthopedic surgery procedures. Energy status energy status and protein intake, nutrition factors known to affect muscle mass and strength in orthopedic patients, has not been characterized prior to admission. Whether this aspect of nutritional status might predict recovery of muscle mass, strength, and function in the context of standard practice/post-operative rehabilitative treatment guidelines is not known.

Elective orthopedic surgery patients face major challenges in maintaining muscle mass and function during the perioperative period. Patients receiving protein or essential amino acid supplementation following total hip and total knee replacement, show improvements in protein balance, patient reported outcome measures, as well as muscle mass, strength, and function. Investigations of larger sample size and longer study duration where protein intake is adequately characterized prior to surgery are needed in these patient populations to further determine connections between routine protein intake and post-operative muscle specific outcomes. Perioperative nutrition screening and assessment measures specifically tailored to orthopedic patients that are attentive to energy status and protein intake are needed. The development and validation of the protein screener proposed in for this project is a unique approach to efficiently acquiring valuable perioperative dietary information. Including subjective, as well as functional, outcome measures may reveal associations between energy status and dietary protein intake pre-operatively and rehabilitative outcomes specific to muscle health to support routine assessment of these dietary factors as prognostic indicators for patient recovery following total hip and total arthroplasty. The proposed project is novel in its goal to establish a foundation for evidence-based rehabilitative nutrition guidelines to enhance perioperative patient care and improve post-operative rehabilitative outcomes specific to muscle health (i.e., strength and function) and quality of life in elective orthopedic surgery patients undergoing total joint replacement procedures.

Approach. Following approval of investigation by the Hartford Hospital Institution Review Board, data collection involved the inclusion of a research information sheet and a 3-day food record with instructions for the respective patient to complete prior to surgery. Recruitment was done in collaboration with the perioperative program staff. Eligible patients and a member of the research team met with patients to determine interest, review study requirements, and obtain written, informed consent for study enrollment. Dietary assessments (protein screener and 3-day food record) occurred before and after surgery per treatment guidelines for total hip and total knee replacement patients, respectively. The protein screener was designed to characterize protein intake and protein source and the respective 3-day food record for participants was used to validate patient responses on screener. Routine clinical assessments per treatment guidelines for respective patient populations were done.

Statistical Approach. Means and standard deviations were determined for outcome measures. Data was analyzed using a 3 factor (energy status, protein intake, and rehabilitative outcome measures) repeated measures over time analysis of variance. Post hoc tests were applied where statistical significance is noted; alpha-level was set at P< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5-34.9 kg/m2; receiving elective total hip or knee arthroplasty due to osteoarthritis for first time

Exclusion Criteria:

* Patients with any non-orthopedic impairment that can impact lower extremity function or mobility, such as paralysis, stroke, multiple sclerosis, and spinal cord injury

Post-enrollment exclusion criteria (if applicable)

For Aim 2:

* Patients who do not attend post-operative physical therapy at one of the identified locations (please see section: Project Personnel)
* Patients who are non-compliant with their physical therapy prescription (missing four or more scheduled sessions).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 50-70 yrs undergoing first elective total joint arthroplasty for hip or knee.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Protein Intake | Protein intake will be assessed 1-2 weeks before surgery and postoperatively at day 1, Week 2, and 6 months for total hip arthroplasty patients
  Protein intake will be determined inadequate (less than 1.2 g/kg/day) or adequate (greater than or equal to 1.2g/kg/day)
Protein Intake | Protein intake will be assessed 1-2 weeks before surgery postoperatively between Day 1 to Week 2, at 4 to 6 Weeks, and at 7 to 12 Weeks for total knee arthroplasty patients
  Protein intake will be determined inadequate (less than 1.2 g/kg/day) or adequate (greater than or equal to 1.2g/kg/day)

SECONDARY OUTCOMES:
Energy balance (i.e., positive or negative balance determined as difference between estimates of calorie/energy intake and energy expenditure) | Energy balance/status will be assessed 1-2 weeks before surgery and postoperatively at day 1, Week 2, and 6 months for total hip arthroplasty patients.
  Energy balance is determined as difference between calories estimated for energy expenditure and calories consumed. Energy intake will be determined from the 3 day food records provide by study participants and energy expenditure will be estimated using the Mifflin-St. Jeor predictive equation plus calories estimated using respective activity factors for participating subjects.
Energy balance (i.e., positive or negative balance determined as difference between estimates of calorie/energy intake and estimates of energy expenditure) | Energy balance/status will be assessed 1-2 weeks before surgery postoperatively between Day 1 to Week 2, at 4 to 6 Weeks, and at 7 to 12 Weeks for total knee arthroplasty patients
  Energy balance is determined as difference between calories estimated for energy expenditure and calories consumed. Energy intake will be determined from the 3 day food records provide by study participants and energy expenditure will be estimated using the Mifflin-St. Jeor predictive equation plus calories estimated using respective activity factors for participating subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Rodriguez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Hartford Hospital Bone & Joint Institute, Hartford, Connecticut, United States

REFERENCES:
- [Background] Mizner RL, Petterson SC, Clements KE, Zeni JA Jr, Irrgang JJ, Snyder-Mackler L. Measuring functional improvement after total knee arthroplasty requires both performance-based and patient-report assessments: a longitudinal analysis of outcomes. J Arthroplasty. 2011 Aug;26(5):728-37. doi: 10.1016/j.arth.2010.06.004. Epub 2010 Sep 20. PMID 20851566
- [Background] Howard EE, Pasiakos SM, Fussell MA, Rodriguez NR. Skeletal Muscle Disuse Atrophy and the Rehabilitative Role of Protein in Recovery from Musculoskeletal Injury. Adv Nutr. 2020 Jul 1;11(4):989-1001. doi: 10.1093/advances/nmaa015. PMID 32167129
- [Background] Howard EE, Margolis LM, Fussell MA, Rios CG, Meisterling EM, Lena CJ, Pasiakos SM, Rodriguez NR. Effect of High-Protein Diets on Integrated Myofibrillar Protein Synthesis before Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Pilot Study. Nutrients. 2022 Jan 27;14(3):563. doi: 10.3390/nu14030563. PMID 35276922
- [Background] Church DD, Schutzler SE, Wolfe RR, Ferrando AA. Perioperative amino acid infusion reestablishes muscle net balance during total hip arthroplasty. Physiol Rep. 2021 Sep;9(18):e15055. doi: 10.14814/phy2.15055. PMID 34558214
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Dreyer HC, Owen EC, Strycker LA, Smolkowski K, Muyskens JB, Kirkpatrick TK, Christie AD, Kuehl KS, Lantz BA, Shah SN, Mohler CG, Jewett BA. Essential Amino Acid Supplementation Mitigates Muscle Atrophy After Total Knee Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. JB JS Open Access. 2018 Jun 4;3(2):e0006. doi: 10.2106/JBJS.OA.18.00006. eCollection 2018 Jun 28. PMID 30280129
- [Background] Dreyer HC, Strycker LA, Senesac HA, Hocker AD, Smolkowski K, Shah SN, Jewett BA. Essential amino acid supplementation in patients following total knee arthroplasty. J Clin Invest. 2013 Nov;123(11):4654-66. doi: 10.1172/JCI70160. Epub 2013 Oct 25. PMID 24135139
- [Background] Kouw IWK, Groen BBL, Smeets JSJ, Kramer IF, van Kranenburg JMX, Nilwik R, Geurts JAP, Ten Broeke RHM, Poeze M, van Loon LJC, Verdijk LB. One Week of Hospitalization Following Elective Hip Surgery Induces Substantial Muscle Atrophy in Older Patients. J Am Med Dir Assoc. 2019 Jan;20(1):35-42. doi: 10.1016/j.jamda.2018.06.018. Epub 2018 Aug 11. PMID 30108034
- [Background] Dutaillis B, Maniar N, Opar DA, Hickey JT, Timmins RG. Lower Limb Muscle Size after Anterior Cruciate Ligament Injury: A Systematic Review and Meta-Analysis. Sports Med. 2021 Jun;51(6):1209-1226. doi: 10.1007/s40279-020-01419-0. Epub 2021 Jan 25. PMID 33492623